CLINICAL TRIAL: NCT05752630
Title: The Relation Between Physical Activity, Sedentary Behaviour, and Cardiometabolic Health in Multiple Sclerosis
Brief Title: Physical Activity, Sedentary Behaviour and Cardiometabolic Health in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Principal Investigator, Hasselt University
Other Study IDs: CAMS
Record Dates: First submitted 2023-02-01; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Physical activity; Sedentary behaviour; Cardiometabolic health; Comorbidities
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control: Healthy controls who engage in sedentary behaviour for more than 9 hours per day. Strata will be used to ensure equal distribution of active and inactive participants (< and > 150min/MVPA/week)
- Persons with MS: Persons suffering from MS who engage in sedentary behaviour for more than 9 hours per day. Strata will be used to ensure equal distribution of active and inactive participants (< and > 150min/MVPA/week)

SUMMARY:
This study evaluates the association between sedentary behaviour, physical activity, and the cardiometabolic health of Multiple Sclerosis via several cardiovascular, metabolic and anthropometric parameters.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune, inflammatory and neurodegenerative disorder of the central nervous system, predominantly affecting young to middle-aged adults. The disease manifests in a broad spectrum of associated sensory, motor and psychological dysfunction, and there is a large variability in symptoms between (and within) persons with MS (PwMS). This can (partly) be explained by the co-existence of cardiometabolic (CM) diseases, such as hypertension, dyslipidaemia, insulin resistance or diabetes. More specifically, the presence of one or more of these CM diseases has been associated with a worsening of disability, independent of the timing of their development (at MS symptom onset, diagnosis, or later in the disease course). Therefore, the prevention and/or treatment of these CM comorbidities also warrant attention in MS rehabilitation.

In most studies PwMS and HC were matched on age, sex, height and weight. Importantly, differences in physical activity (PA) and sedentary behaviour (SB) were never taken into account, while this might be a relevant matching risk factor between groups. Moreover, Ranadive et al. found a significant worse vascular function in PwMS compared to HC, but differences were accounted for by low PA in PwMS. This might mean that PwMS can completely attenuate their increased CM risk by increasing their PA. However, this conclusion was only based on a statistical correction, there was a large difference in PA between groups and other confounding factors (such as PA intensity, smoking and nutrition intake) were not taken into account.

Therefore, the present study aims to investigate the relation between CM health and different intensities of PA and SB in PA-matched PwMS and HC. When CM health is comparable between PwMS and HC with similar PA levels, this shows the importance of including PA and SB measures and interventions as early as possible in MS treatment before automatically starting CM medication because PwMS are known to have multiple risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Relapse-remitting MS
* 25-60 years old
* EDSS < 5
* Sedentary behaviour (>9hours daily)

Exclusion Criteria:

* <9h SB/day,
* experienced an acute exacerbation within 6 months before the start of the study
* an expanded disability status scale (EDSS) score >5
* experimental drug use or medication changes in the last month
* medical conditions precluding PA participation
* alcohol abuse (>20 units/week)
* reported dietary habits or weight loss (>2kg) in the last month before the study
* intention to start a new specific diet or start to follow an exercise intervention
* reported participation in another biomedical trial which may have an effect on blood parameters 1 month before the start of the study
* blood donation in the past month
* diagnosis of cardiometabolic diseases such as diabetes mellitus or heart and vascular diseases.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Persons with and without Multiple Sclerosis (MS), who also engage for more than 9h per day in sedentary behaviour. Healthy controls will be matched with persons with MS based on their physical activity level, gender, age and BMI.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Body weight | After 7 days of physical activity monitoring
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1 kg
Height | After 7 days of physical activity monitoring
  Body height is measured to the nearest 0.1cm using a wall-mounted Harpenden stadiometer, with participants barefoot
DEXA (Dual Energy X-Ray) | After 7 days of physical activity monitoring
  body fat mass and lean tissue mass using Dual Energy X-ray Absorptiometry
Waist circumference | After 7 days of physical activity monitoring
  Waist circumference will be measured to the nearest 0.1cm using a flexible metric measuring tape with participants barefoot (in underwear) in standing position. Waist circumference is measured at the midpoint between the lower rib margin and the top of the iliac crest.
Hip circumference | After 7 days of physical activity monitoring
  Hip circumference will be measured to the nearest 0.1cm using a flexible metric measuring tape with participants barefoot (in underwear) in standing position. Hip circumference is measured at the widest circumference of the hip at the level of the greater trochanter.
Concentration of glucose | After 7 days of physical activity monitoring
  Concentration of glucose measured in blood analysis during OGTT
Concentration of Insulin | After 7 days of physical activity monitoring
  Blood analysis of insulin during OGTT
Concentration of total cholesterol | After 7 days of physical activity monitoring
  Blood analysis
Concentration of high density lipoprotein cholesterol (HDL-cholesterol | After 7 days of physical activity monitoring
  Blood analysis
Concentration of low density lipoprotein cholesterol (LDL-cholesterol) | After 7 days of physical activity monitoring
  Blood analysis
Concentration of triglyceride | After 7 days of physical activity monitoring
  Blood analysis
Concentration of inflammatory markers | After 7 days of physical activity monitoring
  blood analysis of IL-6, TNF-α and C-reactive protein
Reactive hyperaemia index (RHI) | After 7 days of physical activity monitoring
  Vascular endothelial function will be assessed by non-invasive peripheral arterial tonometry using the EndoPAT™ 2000 device. The reactive hyperaemia index reflects the reactive hyperaemia response, and is calculated as the ratio of the average peripheral arterial tone (PAT) signal in the posthyperemic phase to the baseline PAT signal in the occluded arm, with normalization to the ratio of the PAT signal in the control arm to account for any systemic hemodynamic changes.
Homeostatic model assessment for insulin resistance (HOMA-IR) | After 7 days of physical activity monitoring
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity using the homeostatic model assessment for insulin resistance (HOMA-IR). The HOMA-IR is calculated from the fasting insulin and glucose concentration.sensitivity and beta cell function. The following parameters are calculated: homeostatic model assessment for insulin resistance, whole-body insulin sensitivity index, insulinogenic index and the area under the curve for glucose and insulin.
Insulinogenic index | After 7 days of physical activity monitoring
  An oral glucose tolerance test will be performed for assessment of beta cell function by calculation of the insulinogenic index. The insulinogenic index is calculated from both insulin and glucose concentrations.
Area under the curve of glucose and insulin concentrations | After 7 days of physical activity monitoring
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity by calculation of the area under the curve of glucose and insulin concentrations
Cardiac autonomic function | After 7 days of physical activity monitoring
  Cardiac autonomic function will be operationalized as heart rate variability by means of continuous beat-to-beat heart rate signal measurements. time domain and frequency domain analysis of the R-R intervals will be performed
Systolic and Diastolic blood pressure | After 7 days of physical activity monitoring
  Systolic, diastolic and mean arterial blood pressure will be measured 3 times at 5-min intervals using an electronic sphygmomanometer
metabolic syndrome (MetS) risk score | After 7 days of physical activity monitoring
  A continuous metabolic syndrome risk score will be calculated using the waist circumference, HDL concentration, systolic blood pressure, triglycerides and fasting glucose levels, as described by Gurka et al. (2014). A higher score indicates worse health. Because this is a continuous scale, there is no minimum and maximum value.
Oxygen uptake (VO2) | After 7 days of physical activity monitoring
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VO2 is collected breath-by-breath and averaged every ten seconds.
Respiratory gas exchange ratio (RER) | After 7 days of physical activity monitoring
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis RER is collected breath-by-breath and averaged every ten seconds.
Heart rate (HR) | After 7 days of physical activity monitoring
  Cardiopulmonary exercise test on an electronically braked cycle ergometer is performed. With the aid of a heart rate monitor the HR is measured and averaged every ten seconds.
Arterial stiffness | After 7 days of physical activity monitoring
  Arterial stiffness will be determined by pulse wave analysis (PWA) and pulse wave velocity (PWV) using SphygmoCor (v9; Atcor Medical).
Whole-body insulin sensitivity (WBISI) | After 7 days of physical activity monitoring
  (fasting) glucose and (fasting) insulin levels measured during blood analysis from OGTT are used to calculate whole body-insulin sensitivity.

SECONDARY OUTCOMES:
Steps per day | 7 days
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | 7 days
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | 7 days
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Walking time | 7 days
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sleeping time | 7 days
  Participants will have to keep track of their sleeping time by means of a sleep diary
Exercise information | 7 days
  Participants will have to keep track of their exercise information by means of a diary
Total calorie intake | 7 days
  Participants will record all food and beverages consumed over seven consecutive days and from this the total calorie intake is calculated.
Macronutrient content | 7 days
  Participants will record all food and beverages consumed over seven consecutive days and from this the macronutrient content is calculated.
12-Item Multiple Sclerosis Walking Scale (MSWS-12) questionnaire | After 7 days of physical activity monitoring
  The MSWS-12 is a 12-item patient-rated measure of the impact of MS on walking over the past 2 weeks. The items are rated on a 5-point scale from 1 (Not at all) to 5 (Extremely).
RAND-36 Item Health Survey (RAND-36) questionnaire | After 7 days of physical activity monitoring
  The RAND-36 (RAND refers to the American research organisation that developed the questionnaire; Research And Development') is a generic health profile that consists of two summary scales: a physical component summary (PCS) and a mental component summary (MCS). The total score is transformed to a hundred point scale. A higher score indicates a better health condition
Modified fatigue impact scale (MFIS) questionnaire | After 7 days of physical activity monitoring
  The perceived impact of fatigue on physical, cognitive and psychosocial functioning of the past 4 weeks is assessed in the MFIS. A higher score indicates higher fatigue. The minimum and maximum value for the physical subscale is 0-36, for the cognitive subscale 0-40 and for the psychosocial subscale 0-8, resulting in a total score ranging from 0 to 84.
Perceived stress scale (PSS) questionnaire | After 7 days of physical activity monitoring
  The PSS measures the level to which a respondent considers his or her life stressful and was designed to assess how unpredictable and controllable a person appraises his or her life. The PSS consists of 14 items ranging from 0 to 4. The total score is summed, a higher score indicates more stress.

CONTACTS AND LOCATIONS:
Overall Officials: Bert Op 't Eijnde, prof.dr., Study Chair — Hasselt University; Ine Nieste, drs., Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium